CLINICAL TRIAL: NCT03188549
Title: Magen Haim Project - Assessing Hand Hygiene Formulas
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-17-3882-GR-CTIL
Record Dates: First submitted 2017-05-29; First posted 2017-06-15 (Actual); Last update posted 2017-10-17 (Actual); Status verified 2017-06

CONDITIONS: Comparing Use of Hand Hygiene Products
MeSH Terms: interventions — Clioquinol

STUDY DESIGN:
Intervention Model Description: Comparative research, Cross-Over, with a quasi-experimental component, comparing trial products to the use of Septol over the course of the year before the research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Departments of Branch A (Active Comparator): Intervention: AniosGel Respiratory ICU Pediatric Cardiac Surgery, NICU Hemato-Oncology, Oncology Internal A, C, D, E, F Surgery C, Vascular Surgery and Chest Surgery Pediatric B South Imaging Orthopedics B
  Interventions: Other: AniosGel 85 NPC
- Departments of Branch B (Active Comparator): Intervention: Softaman Neurosurgery ICU Cardiac Surgery, Cardiac ICU, Pediatric ICU Pediatric Hemato-Oncology Internal B and I, Geriatric C and D Surgery B Pediatric B North Emergency Room Orthopedics A and Hand
  Interventions: Other: Softa-Man (Braun)
- Branch C (Active Comparator): Control Intervention - Septol without any changes All patients hospitalized in the 29 departments in Sheba, including two of the branches, during the year of the study
  Interventions: Other: Septol

INTERVENTIONS:
Other: AniosGel 85 NPC — Hand hygiene formula
  Arms: Departments of Branch A
Other: Softa-Man (Braun) — Hand hygiene formula
  Arms: Departments of Branch B
Other: Septol — alcohol-based hand rub
  Arms: Branch C

SUMMARY:
Background: Procedures of hand hygiene are an important component in prevention of cross-transmission of infections in hospitals. In recent years, hand washing with antiseptic soap (chlorhexidine) was replaced with use of alcohol-based hand rub. This change brought an increase in compliance with hand hygiene regulations from 30-40% to over 50%, and in other places up to 70%. However, even 70% compliance is not enough. One of the reported reasons for lack of compliance of staff to the use of alcohol-based preparations is skin irritation and dryness of the hands as a result of frequent use. At Sheba, like the majority of Israeli hospitals, the product used for handwashing is Septol (Teva), which includes 0.5% chlorhexidine gluconate (CHG) and 70% ethyl alcohol. The CDC, WHO and FDA guidelines approve for use of hospital hand hygiene, products that contain between 61-85% ethanol.

The investigators will replace the Septol currently used with a different alcohol-based antiseptic that is more user-friendly, and aim to determine whether this will increase the compliance with hand hygiene protocols.

The investigators will assess

1. Satisfaction of staff.
2. Increase of hand hygiene compliance.

DETAILED DESCRIPTION:
RESEARCH PATTERN:

Comparative research, Cross-Over, with a quasi-experimental component, comparing trial products to the use of Septol over the course of the year before the research.

Included in the study will be 29 departments of Sheba, whilst the other hospital departments will serve as a control group. The 29 departments will be divided into two branches with similar departments in each (each branch consisting of 3 internal medicine departments, 3 urgent care departments, a pediatric department, a surgical department, etc.). In Stage I (the initial six months), Branch A will exchange Septol with AniosGel, and Branch B will exchange Septol with Softa-Man. In Stage II (the second six months), Branch A will change to Softa-Man and Branch B will change to AniosGel. Branch C will be the control, where Septol will be used throughout the duration of the study.

STUDY POPULATION:

For objectives 1 and 2: All medical staff at Sheba (in all 3 branches of the study).

Total: 15 Departments in Branch A, 14 Departments in Branch B

Stages of the Study:

1. At point zero (while still using Septol), distribute a questionnaire of hand hygiene compliance and satisfaction.
2. Instruction to Branch A and Branch B departments regarding the switch of Septol to the new product (instruction to staff in all sectors of these departments).
3. Exchange antiseptic Septol with the trial product in departments of Branch A and Branch B for the first six months (Stage I).
4. At point one (six months into the study), distribute a questionnaire of hand hygiene compliance and satisfaction.
5. Interim analysis of the questionnaires from point zero and point one.
6. Instruction to departments regarding the switch of products, regarding the use of the new product.
7. Exchange of trial product between the two groups for the second six month period (Stage II).
8. At point two (twelve months into the study), distribute a questionnaire of hand hygiene compliance and satisfaction.
9. Final analysis of questionnaires from Point 0, 1, and 2, as well as compliance of hand hygiene.

ELIGIBILITY:
Inclusion Criteria:

* All staff in the participating departments

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1505 (Estimated)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-06-15 (Estimated); Study Completion 2019-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of staff reporting satisfaction with hand hygiene formula in questionnaire | 1 year
  Satisfaction Questionnaire will be distributed and filled in three times during the study.
Percentage of proper hand hygiene compliance as determined by Chess Application | 1 year
  The Chess Program, an application designed for analyzing compliance, will be used by researchers to observe and record amounts of times that staff members comply or do not comply with proper hand hygiene protocols, and determine the percentage of times that staff complied with proper hand hygiene protocols out of all observations

SECONDARY OUTCOMES:
Hand Hygiene Formula Use | 1 year
  Measuring the amount of product used, amount of bottles per hospitalization bed according to department (an accepted surrogate model measurement of hand hygiene compliance).

CONTACTS AND LOCATIONS:
Overall Officials: Dror Harats, Prof., Study Chair — IRB Committee Sheba Medical Center Israel
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No